CLINICAL TRIAL: NCT02776098
Title: Muscle Accrual and Function in Cystic Fibrosis-Impact of Glucose Intolerance
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of Pennsylvania (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 15-012279; 1K23DK107937-01 (NIH)
Record Dates: First submitted 2016-05-16; First posted 2016-05-18 (Estimated); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Glucose Intolerance; Muscle Accrual; Cystic Fibrosis-related Diabetes; Healthy Controls; Healthy Participants
MeSH Terms: conditions — Cystic Fibrosis; Glucose Intolerance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Cystic Fibrosis without Cystic Fibrosis-related Diabetes: Subjects with a confirmed diagnosis of Cystic Fibrosis (CF) without Cystic Fibrosis-related diabetes will be followed annually for 2 years for a total of four study visits over 2 years (screening, baseline, 12 and 24 month visits).
- Newly Diagnosed Cystic Fibrosis-Related Diabetes: Subjects with a confirmed diagnosis of Cystic Fibrosis (CF) and new diagnosis of Cystic Fibrosis-Related Diabetes (CFRD) will be followed for a total of 3 study visits over 6 months (screening, baseline and 6 months).
- Healthy Controls: Age, sex, ethnicity and body mass index matched (at time of enrollment to CF without CFRD subjects) healthy controls will be followed annually for 2 years for a total of four study visits (screening, baseline, 12 and 24 month visits).

SUMMARY:
This study will investigate the link between glucose abnormalities and elements critical to muscle function including mass, composition and energy metabolism. the primary goal of the study is to determine whether Cystic Fibrosis (CF) disease is associated with muscle dysfunction, especially in the presence of glucose intolerance. This is a longitudinal cohort study of 3 main groups: CF subjects without Cystic Fibrosis-related diabetes (CFRD), healthy matched controls and CF subjects with newly diagnosed CFRD started on insulin therapy.

DETAILED DESCRIPTION:
Cystic Fibrosis (CF) is a lethal inherited disease that primarily affects the lungs but also confers a high risk of diabetes, with up to 40-50% of adults experiencing Cystic Fibrosis-related diabetes (CFRD). CFRD is associated with an accelerated decline in lung function, nutritional status and survival and despite treatment mortality in patients with CFRD remains high. Airway inflammation and susceptibility to infections caused by hyperglycemia, and the catabolic effect of insulin deficiency are posited mechanisms of CFRD-associated morbidity. Respiratory failure caused by airway disease is well known but the contribution of respiratory muscle dysfunction may be critical. In Type 2 Diabetes Mellitus (T2DM) glucose and insulin defects are closely correlated with muscle function. The pulmonary muscles are crucial to respiration and airway clearance in CF. Muscle function is dependent on its mass, composition, and energy metabolism. Lean body mass (LBM) deficits are present in CF and improvement in LBM improves pulmonary function. Using T2DM as a model for muscle dysfunction, the study hypothesis is that glucose intolerance exacerbates LBM deficits, negatively affects muscle composition, and alters muscle metabolism leading to respiratory muscle dysfunction and a decline in pulmonary function.

CF subjects without CFRD and healthy controls will undergo 3 study visits (baseline then annually for 2 years) and CFRD subjects will undergo 2 study visits (baseline and 6 months after baseline). Evaluations will include neurologic exams, anthropometric assessments, 3-day dietary recall, MRI scans, oral glucose tolerance tests (CF subjects only), blood work, pulmonary function testing, muscle strength testing, exercise testing, bone density scans, and adverse event assessment.

ELIGIBILITY:
Inclusion Criteria for CF subjects without CFRD:

1. Males or females age 16 to 22 years.
2. Confirmed diagnosis of CF per CF Foundation guidelines
3. Parental/guardian permission (informed consent) and if appropriate, child assent.

Exclusion Criteria for CF subjects without CFRD

1. Chronic systemic glucocorticoid use e.g. for allergic bronchopulmonary aspergillosis
2. Organ transplantation
3. Forced Expiratory Volume (FFEV) 1%-predicted < 40%
4. Established diagnosis of CFRD and treatment with insulin or hypoglycemic agent
5. Parents/guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.
6. Pregnancy or breastfeeding (if female)
7. Pre-existing neurological or neuromuscular disease

All study visits for CF subjects will be scheduled during periods of baseline health. Visits will not be performed within 4 weeks of an acute respiratory illness or pulmonary exacerbation.

Inclusion Criteria for healthy controls

1. Age-, sex-, ethnicity-, and BMI-matched at time of enrollment to CF subjects without CFRD
2. Parental/guardian permission (informed consent) and if appropriate, child assent.

Exclusion Criteria for healthy controls

1. Parents/guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.
2. Pregnancy or breastfeeding (if female)
3. Pre-existing neurological or neuromuscular disease

Inclusion Criteria for CF subjects with new CFRD

1. Males or females age 12 years or above.
2. Confirmed diagnosis of CF per CF Foundation guidelines.
3. New diagnosis of CFRD based on a) a clinically indicated Oral glucose tolerance test (OGTT) b) hyperglycemia (PG>200 mg/dL) persisting >48 hours and/or c) elevated HbA1C and within 4 weeks of starting insulin therapy.
4. Parental/guardian permission (informed consent) and if appropriate, child assent.

Exclusion Criteria for CF subjects with new CFRD

1. Chronic systemic glucocorticoid use e.g. for allergic bronchopulmonary aspergillosis
2. Organ transplantation
3. Parents/guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.
4. Pregnancy or breastfeeding (if female)
5. Pre-existing neurological or neuromuscular disease

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This is longitudinal cohort study of 3 main study groups: CF subjects without CFRD, Healthy matched controls and CF subjects with newly diagnosed CFRD started on insulin therapy. Healthy controls without CF will be recruited and will be matched for age, sex, ethnicity, and body mass index (BMI) to CF subjects. Subjects with newly diagnosed CFRD will also be enrolled. This study will be carried out over a 5-year period.
  CF subjects without CFRD (26) and healthy controls (26) will be followed annually for 2 years. CF subjects with newly diagnosed CFRD (10) will be followed for 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2016-05; Primary Completion 2024-03-04 (Actual); Study Completion 2024-03-04 (Actual)

PRIMARY OUTCOMES:
Compare change in mean lean body mass (LBM) from baseline to end of study | 24 months (CF without CFRD subjects & healthy controls); 6 months for CF subjects

SECONDARY OUTCOMES:
Compare Intramyocellular lipid (IMCL) accumulation from baseline to end of study | 24 months (CF without CFRD subjects & healthy controls); 6 months for CF subjects
  Proton magnetic resonance spectroscopy will be used to measure IMCL per previously published methods.

CONTACTS AND LOCATIONS:
Overall Officials: Clement L Ren, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (2):
- United States (2):
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No